CLINICAL TRIAL: NCT03994393
Title: A Phase 2 Trial of Durvalumab (MEDI4736) and Tremelimumab With Chemotherapy in Metastatic EGFR Mutant Non-squamous Non-small Cell Lung Cancer (NSCLC) Following Progression on EGFR Tyrosine Kinase Inhibitors (TKIs)
Brief Title: Non Small Cell Lung Cancer Trial of Durvalumab and Tremelimumab in Advanced Epidermal Growth Factor Receptor (EGFR) Mutant Disease.
Acronym: ILLUMINATE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sydney (Other)
Collaborators: AstraZeneca (Industry); Australasian Lung Cancer Trials Group (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTC 0209; ALTG 16/009 (Other: The Australasian Lung Cancer Trials Group)
Record Dates: First submitted 2019-06-20; First posted 2019-06-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: EGFR Mutant Advanced Non Small Cell Lung Cancer
MeSH Terms: interventions — tremelimumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Active Comparator): Participants with no evidence of T790M
  Interventions: Drug: Tremelimumab; Drug: Durvalumab
- Cohort 2 (Active Comparator): Participants with evidence of T790M
  Interventions: Drug: Tremelimumab; Drug: Durvalumab

INTERVENTIONS:
Drug: Tremelimumab — During induction, patients will receive 4 cycles of durvalumab 1500mg and tremelimumab 75mg with cisplatin 75mg/m2 (or carboplatin AUC 5 if cisplatin is contra-indicated), and pemetrexed 500mg/m2 via intravenous infusion every 3 weeks.
  Followed immediately by a maintenance phase of durvalumab 1500mg and pemetrexed 500mg/m2 once every 4 weeks via intravenous infusion until disease progression or intolerance.
Drug: Durvalumab — During induction, patients will receive 4 cycles of durvalumab 1500mg and tremelimumab 75mg with cisplatin 75mg/m2 (or carboplatin AUC 5 if cisplatin is contra-indicated), and pemetrexed 500mg/m2 via intravenous infusion every 3 weeks.
  Followed immediately by a maintenance phase of durvalumab 1500mg and pemetrexed 500mg/m2 once every 4 weeks via intravenous infusion until disease progression or intolerance.

SUMMARY:
The primary purpose of this trial is to evaluate the efficacy and tolerability of durvalumab and tremelimumab with platinum-pemetrexed in patients with metastatic NSCLC (T790+ve or T790M-ve) following progression on EGFR Tyrosine Kinase Inhibitors..

Study population:

Individuals may be eligible to enrol in this trial if aged 18 or over and have been diagnosed with advanced non-small cell lung cancer (T790+ve or T790M-ve) following progression on EGFR Tyrosine Kinase Inhibitors.

Study details:

All participants enrolled in this trial will begin with induction therapy which involves 4 cycles of durvalumab 1500mg and tremelimumab 75mg with cisplatin 75mg/m2 or carboplatin AUC 5, and pemetrexed 500mg/m2 intravenously every 3 weeks.

Participants will then move into a maintenance phase of durvalumab 1500mg and pemetrexed 500mg/m2 once every 4 weeks until disease progression or unacceptable side effects.

All patients will be reviewed every three to four weeks by blood samples, CT scans and side effect assessments.

It is hoped that the findings from this trial will provide information on whether treatment with durvalumab and tremelimumab with platinum-pemetrexed is feasible, safe and effective for the treatment of advanced non-small cell lung cancer (T790+ve or T790M-ve).

ELIGIBILITY:
Inclusion Criteria:

1. Adults, aged 18 years and older with histologically and/or cytologically confirmed non-squamous non-small cell lung cancer with EGFR mutation of Exon 19 deletion or Exon 21 L858R point mutation.

   * Patients with co-mutations are allowed as long as one of the mutation is either Exon 19 deletion or Exon 21 L858R point mutation
   * Patients with mixed histology must have non-squamous NSCLC as the predominant histology.
2. Disease that has progressed and either:

   (i) No evidence of EGFR T790M resistance mutation in both tissue re-biopsy and plasma after one-line of EGFR tyrosine kinase inhibitor therapy (TKI) OR (ii) T790M mutation (detected in tissue re-biopsy, plasma or both) and progression on 3rd generation EGFR TKI; patients are allowed to have one prior line of TKI therapy before 3rd generation TKI
3. Measurable disease according to RECIST 1.1
4. ECOG performance status of 0 or 1
5. Adequate bone marrow function as defined below (within 14 days prior to registration and with values within the ranges specified below):

   * Platelets equal to or greater than 100 x 109/L
   * Absolute neutrophil count (ANC) equal to or greater than 1.0 x 109/L (equal to or greater than 1000 per mm3)
   * Haemoglobin equal to or greater than 90 x g/L
6. Adequate liver function (within 14 days prior to registration and with values within the ranges specified below):

   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) equal to or less than 2.5 x institutional upper limit of normal (ULN). (or equal to or less than 5 x ULN if liver metastases are present)
   * Bilirubin equal to or less than 1.5 x ULN
7. Adequate renal function (within 14 days prior to registration):

   • Measured creatinine clearance greater than 40 mL/min or Calculated creatinine clearance greater than 40 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine clearance
8. Provision of a pre-treatment tumour tissue sample from a biopsy taken within 42 days prior to enrolment (core biopsy preferred) to determine NSCLC histology and for translational research.
9. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients.
10. Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
11. Signed written informed consent (main study and optional biobanking).

Exclusion Criteria:

1. Prior chemotherapy or immunotherapy, including prior anti-PD-1/anti-PD-L1 or anti-CTLA-4 antibodies, for advanced NSCLC.

   * For recurrent, incurable disease, prior adjuvant chemotherapy or concurrent chemotherapy and radiotherapy with curative intent is allowed, but must have been completed more than 6 months ago, and must not have included treatment with an immune checkpoint inhibitor.
   * Prior EGFR-TKI (e.g. erlotinib, gefitinib, afatinib or osimertinib), including experimental TKI agents, within 8 days or approximately 5 x half-life, whichever is the longer, of the first dose of study treatment is allowed. (If sufficient washout time has not occurred due to schedule or PK properties, an alternative appropriate washout time based on known duration and time to reversibility of drug related adverse events could be agreed upon by contacting the ILLUMINATE Study Team).
2. Mixed histology with any small cell or squamous component.
3. Life expectancy of less than 3 months.
4. Current enrolment or participation in another clinical study with an investigational product during the last 12 months, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study must first be discussed with ILLUMINATE Study Team before study enrolment.
5. Any unresolved toxicity NCI CTCAE equal to or greater than Grade 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

   * Patients with equal to or greater than Grade 2 neuropathy will be evaluated on a case-by-case basis after consultation with the ILLUMINATE Study Team.
   * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the ILLUMINATE Study Team.
6. Radiotherapy or major surgery (as defined by the local investigator) within 4 weeks of the first dose of study drug. Note: Local surgery on isolated lesions for palliative intent is acceptable.
7. History of pneumonitis or pulmonary fibrosis with clinically significant impairment of pulmonary function.
8. History of active primary immunodeficiency or allogeneic transplant.
9. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis (with the exception of diverticulosis), systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

   * Patients with vitiligo or alopecia
   * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
   * Any chronic skin condition that does not require systemic therapy
   * Patients without active disease in the last 5 years may be included but only after consultation with the study physician
   * Patients with celiac disease controlled by diet alone
10. Concurrent illness, including severe infection that may jeopardise the ability of the patient to undergo the procedures outlined in this protocol with reasonable safety.
11. History of another primary malignancy except for

    * Malignancy treated with curative intent and with no known active disease equal to or greater than 5 years before the first dose of IP and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    * Adequately treated carcinoma insitu without evidence of disease.
12. Any history of leptomeningeal carcinomatosis, or untreated central nervous system metastases obtained during the screening period or identified prior to signing the PICF. Patients whose brain metastases have been treated may participate provided they show radiographic stability (defined as disease stability on imaging 4 weeks after commencing radiotherapy). Any neurologic symptoms that developed either as a result of the brain metastases or their treatment must have resolved or be stable either, without the use of steroids, or are stable on a steroid dose of equal to or less than 10mg/day of prednisone or its equivalent (and anti-epileptic drugs) for at least 14 days prior to the start of treatment.
13. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
14. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab or tremelimumab. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical steroids, or local steroid injections (e.g. intra articular injection)
    * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    * Steroids as premedication for hypersensitivity reactions (e.g. CT scan premedication)
15. Live attenuated vaccine within 30 days prior to the first dose of study drug, whilst receiving study drug and up to 30 days after the last dose of study drug.
16. Serious medical or psychiatric conditions that might limit the ability of the patient to comply with the protocol.
17. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab plus tremelimumab combination therapy.
18. Known allergy or hypersensitivity to any of the study drugs or excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Objective tumour response rate (OTRR) and Objective tumour response (OTR) | 36 months post enrolment of first participant.
  Objective tumour response rate (OTRR) as defined by RECIST 1.1. Objective tumour response (OTR) is defined as a partial response or compete response by RECIST 1.1. OTRR is defined as the proportion (percentage) of participants with a confirmed CR or PR according to RECIST 1.1.

SECONDARY OUTCOMES:
Disease control (Disease Control Rate (DCR) | 36 months post enrolment of first participant.
  Disease control (Disease Control Rate (DCR) = Complete Response (CR) + Partial Response (PR) + Stable Disease (SD) as defined by RECIST 1.1.
Objective tumour response rate (OTRR) & Objective tumour response (OTR) | 36 months post enrolment of first participant.
  Objective tumour response rate (OTRR) as defined by iRECIST. Objective tumour response (OTR) is defined as a partial response or compete response by iRECIST. OTRR is defined as the proportion (percentage) of participants with a confirmed CR or PR according to iRECIST.
Progression-free survival (PFS) | 36 months post enrolment of first participant.
  Progression-free survival (PFS) as defined by RECIST 1.1 and iRECIST. PFS is defined as the interval from date of registration to the date of first evidence of disease progression or death, whichever occurs first. Disease progression is defined according to RECIST 1.1 and iRECIST.
Progression-free survival at 12 months (PFS12) | 12 months post enrolment of last participant.
  Progression-free survival at 12 months (PFS12) as defined by RECIST 1.1 and iRECIST. PFS at 12 months taken to mean 1 calendar year, i.e. 365 days. Study participants who have stable disease, partial response or complete response confirmed at the first scheduled assessment after 12 months according to RECIST v1.1 will be considered to have attained PFS at 12 months.
Overall survival (OS) | 36 months from enrolment of first participant.
  Overall survival (OS) is defined as the interval from the date of registration to date of death from any cause, or the date of last known follow-up alive.
Number and Severity (assessed as a composite) of Adverse Events | 36 months post enrolment of first participant.
  Number and Severity (assessed as a composite) of Adverse Events - using the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Chee K Lee, Study Chair — St George Hospital, Australia
Locations (16):
- Australia (9):
  - St George Hospital, Kogarah, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Medical Centre - Clayton, Clayton, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - St Vincent's Hospital (Melbourne), Melbourne, Victoria
- Taiwan (7):
  - Taiwan Dalin Tzu Chi Hospital, Chiayi City
  - Taiwan China Medical University Hospital, Taichung
  - Taiwan Taichung Veterans General Hospital, Taichung
  - Taiwan National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taiwan Taipei Veterans General Hospital, Taipei
  - Taiwan Tri-Service General Hospital, Taipei

REFERENCES:
- [Derived] Lee CK, Liao BC, Subramaniam S, Chiu CH, Mersiades AJ, Ho CC, Brown C, Lai CL, Hughes BGM, Yang TY, O'Byrne K, Luo YH, Yip S, Ho CL, Bray V, Su WC, Moore M, Feng WL, Bai YY, Ford K, Cummins MM, Stockler MR, Solomon BJ, John T, Chih-Hsin Yang J. Durvalumab, Tremelimumab, and Platinum Chemotherapy in EGFR Mutation-Positive NSCLC: An Open-Label Phase 2 Trial (ILLUMINATE). JTO Clin Res Rep. 2024 Nov 22;6(2):100771. doi: 10.1016/j.jtocrr.2024.100771. eCollection 2025 Feb. PMID 39877028